CLINICAL TRIAL: NCT06271109
Title: Short Term Surgical Outcomes of Anatomical Versus Non Anatomical Laparoscopic Liver Resection for Liver Tumors
Status: Enrolling by invitation | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amir Ayman Mohamed, principle investigator, Sohag University
Other Study IDs: Soh-Med-24-01-04MD
Record Dates: First submitted 2024-02-05; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Liver Neoplasms
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic Anatomical liver resection
  Interventions: Procedure: Anatomical laparoscopic liver resection for liver neoplasms
- laparoscopic Non Anatomical liver resection
  Interventions: Procedure: Non-Anatomical laparoscopic liver resection for liver neoplasms

INTERVENTIONS:
Procedure: Anatomical laparoscopic liver resection for liver neoplasms — resection of liver tumors laparoscopically based on surgical anatomical segmentation of the liver
  Groups: laparoscopic Anatomical liver resection
Procedure: Non-Anatomical laparoscopic liver resection for liver neoplasms — resection of liver tumors laparoscopically not based on surgical anatomical segmentation of the liver
  Groups: laparoscopic Non Anatomical liver resection

SUMMARY:
aimed to discuss the short term surgical outcomes of Anatomical versus Non anatomical laparoscopic Liver resection for Liver tumors.

DETAILED DESCRIPTION:
This study aimed to be both prospective and retrospective study including the cases of laparoscopic liver resection that was done and will be done during the period from December 2021 to June 2025. This study will include cohort of patients who met the eligible criteria.

Complete history taking with special concern to the following:

* Age, sex and life style.
* present medical history: hepatic condition and other debilitating diseases.
* Past medical History: blood transfusion, hepatitis, liver cirrhosis and history of hospital admission.

Complete local examination of the abdomen including:

* Local examination of the skin overlying for any signs of infection, radiation fibrosis and or presence of sinuses
* Percussion for presence of ascites
* Palpation for cirrhosis or any palpable masses investigations will be carried

  1. Ultrasonography: routine abdominal US for every case.
  2. Triphasic CT scan
  3. CT volumetric study to evaluate remaining liver volume when needed.
  4. Dynamic or triphasic MRI if needed
  5. Metastatic work up (CT chest, bone scan and PET scan in selected patients).
  6. Preoperative histopathological examination when needed.
  7. routine laboratory investigations

ELIGIBILITY:
Inclusion Criteria:

* all patients diagnosed with liver tumors (benign and malignant) lesions suitable for laparoscopic liver resection (Anatomical and Non anatomical)
* Patients with Child Pugh A and early B
* Patients Fit for surgery as regard anesthesia
* Patients who accept to participate in the study and sign an informed consent

Exclusion Criteria:

* Patients with Child Pugh late B&C liver disease.
* For Patients with hepatocellular carcinoma BCLC stage C&D (extra hepatic spread and macro vascular invasion)
* Patients with contraindications to laparoscopic surgery and (or) unfit for surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with liver neoplasms candidate for resection and fit for surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
complete resection of the neoplasm | 3.5 years
  to ensure complete resection with free resection margins

SECONDARY OUTCOMES:
residual liver tissue | 3.5 years
  to evaluate the remnant liver tissue post neoplasm resection
recurrence rate | 3.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt